CLINICAL TRIAL: NCT06147076
Title: Journey to Transplant: Virtual Coaching for Potential Kidney Transplant Patients and Their Social Support Networks
Brief Title: Social Support Counseling Intervention for Kidney Transplant Candidates
Acronym: JtT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01DK135730-01 (NIH)
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant
Keywords: Interventional Counseling; Kidney Transplant; Interventional Mapping; Counseling; Social Support Networks; Dialysis

STUDY DESIGN:
Intervention Model Description: Control group versus interventional group. Questionnaire completed by interventional group and their social support networks pre and post.
Who Masked: Outcomes Assessor
Masking Description: Statisticians will be blinded to group assignment when assessing outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Pre-Transplant Counseling Intervention (No Intervention): Participants in control arm will undergo usual pre-transplant counseling as per the standard of care.
- Social Support Network Counseling Intervention (Experimental): Participants in the intervention arm will undergo an additional pretransplant counseling session along with members of their social support networks after their initial transplant evaluation and counseling.
  Interventions: Behavioral: Social Support Network Counseling Intervention

INTERVENTIONS:
Behavioral: Social Support Network Counseling Intervention — Social support counseling intervention for kidney transplant candidates along with their social support networks.
  Arms: Social Support Network Counseling Intervention

SUMMARY:
Virtual Coaching for Potential Kidney Transplant Patients

DETAILED DESCRIPTION:
Individuals who are eligible for kidney transplant will be recruited by phone or email and randomized into two groups, control and interventional counseling. The control group will be given a simple survey to fill and return while the interventional counseling will go through a group education and counseling session along with members of their social support networks. The interventional counseling will then complete a pre and post survey (same as control group). Survey answers will be recorded within REDCAP.

ELIGIBILITY:
Inclusion

* Determined by transplant center to be suitable for continuation in evaluation for listing (or a member of that person's social support network)
* 18 Years of age or older
* English-speaking
* Willingness to participate with at least 2 social network members in the session and have calculator results shown to social network members (if a patient)
* Able to provide informed consent

Exclusion

* Prisoners
* Individuals with impaired ability to consent
* Pregnant females.
* Patients who choose to opt out of research.
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Correct Answers on Knowledge of Kidney Transplant Options Assessment | one month
  Questionnaire

SECONDARY OUTCOMES:
Decisional Conflict Scores | one month
  Questionnaire
Social Support Scores | one month
  Questionnaire
Knowledge Scores | one month
  Questionnaire
Hearth Hope Index | one month
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin Healthcare, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
There might be an exchange of data with our collaborators with the study at the University of Minnesota-Twin Cities

REFERENCES:
- See also: American Transplant Congress oral abstract — http://atcmeetingabstracts.com/abstract/journey-to-transplant-a-pilot-feasibility-trial-of-a-virtual-counseling-intervention-for-patients-and-their-social-support-networks-to-improve-access-to-kidney-transplant/